CLINICAL TRIAL: NCT03949179
Title: Optimizing Management of Low Back Pain Through the Pain and Disability Drivers Management Model: Study Protocol for a Feasibility Trial
Brief Title: Optimizing Management of Low Back Pain Through the Pain and Disability Drivers Management Model
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: Quebec Pain Research Network (Other)
Responsible Party: Sponsor
Other Study IDs: MP-31-2019-3131
Record Dates: First submitted 2019-04-29; First posted 2019-05-14 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Mechanical Low Back Pain
Keywords: Low back pain; Pain management; Rehabilitation; Feasibility outcomes
MeSH Terms: conditions — Low Back Pain; Agnosia | interventions — Models, Biological

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pain and Disability Drivers Management model: Participating clinicians will use the PDDM model to guide assessment and treatment of their patients for a 6-weeks period.
  Interventions: Device: The Low Back Pain and Disability Drivers Management (PDDM) model

INTERVENTIONS:
Device: The Low Back Pain and Disability Drivers Management (PDDM) model — The Low Back Pain and Disability Drivers Management (PDDM) model aims to identify the domains influencing pain and disability to guide clinical decisions. The model is composed of five domains upon which the clinician can base his assessment and orientate treatment allocation and includes: 1) nociceptive pain drivers (i.e., somatic, inflammatory or mixed pain), 2) nervous system dysfunction (NSD) drivers (i.e., sensitization of the peripheral and/or central nervous system), 3) comorbidity drivers (i.e., physical and/or mental health comorbidities), 4) cognitive-emotional drivers (i.e., maladaptive cognitions and/or behaviors) and 5) contextual drivers (i.e., occupational-related and social environmental contextual drivers). This profiling will inform and lead the clinician's treatment approach based on the combined contribution of each domain driving the experience of pain and disability.

SUMMARY:
This study aims to determine the feasibility of conducting a future randomized controlled trial to collect preliminary data on the effectiveness of a previously validated approach that takes into account all the pain and disability vectors associated with low back pain - the Pain and Disability Drivers Management Model (PDDM).

The overall objective is to provide data to assess the feasibility of implementing a future randomized clinical trial to evaluate the impact of the PDDM on the management of non-specific LBP in a clinical setting and to explore the short-term effect of using the model on patient's clinical outcomes.

DETAILED DESCRIPTION:
Background: Non-specific mechanical low back pain (LBP) is highly prevalent, recurrent and is a leading cause of disability worldwide. Despite increased efforts in improving care, the self-reported levels of disability in individuals with LBP have not improved in the last decade. In order to more effectively manage LBP through non-pharmacological approaches, evidence endorses the use of classification systems to support diagnosis and guide treatments. However, this approach to care is not without limitations and a more comprehensive and broader perspective is needed. Hence, we recently proposed and validated the Low Back Pain and Disability Drivers Management (PDDM) model, which aims to identify the domains influencing pain and disability to create a profile or phenotype to guide clinical decisions. The objective of this study is to assess the feasibility of conducting a trial and to gather preliminary effect outcomes of the intervention in clinical setting.

Methods: The design is a prospective single arm experimental design. Physiotherapists (PTs) working with a population suffering from musculoskeletal disorders and patients presenting with non-specific mechanical LBP from two different clinical settings will be recruited. The intervention consists of a one-day training workshop for PTs on using the PDDM to guide management decisions. PTs will then perform a 6-weeks follow-up with their participating patients. This feasibility study will assess recruitment and retention rates as well as PTs' acceptability and patients' satisfaction outcomes related to the intervention. Preliminary effect outcomes will also be gathered.

Discussion: This study will inform the feasibility and acceptability of the intervention and gather preliminary outcomes to conduct a future randomized controlled trial to measure the effectiveness of the intervention in managing non-specific mechanical LBP.

ELIGIBILITY:
Inclusion Criteria:

Clinicians:

* be working with a population suffering from musculoskeletal disorders such as LBP and have a valid license to practice physiotherapy in the province of Quebec
* agree to participate to the one-day training workshop (intervention)
* assess and initiate treatment of their patients presenting with non-specific LBP guided by our newly developed model

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients:
  * Patients presenting with non-specific LBP according to the assessment conducted by the PT
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of implementation | T1: clinician's baseline.
  Recruitment rate: % of eligible clinicians who enrolled in the study (T1)
Feasibility of implementation | T1: clinician's baseline; T3 (6 weeks)
  Retention rate: % of contacted clinicians who accepted to participate and report data (T3-T1)
Clinician's acceptability of the workshop | T1: clinician's baseline (after the workshop)
  Assessed via semi-structured phone interviews. It includes the clinician's appreciation of the training.
Clinician's acceptability of the intervention | T3 (6 weeks)
  Assessed via semi-structured phone interviews and include clinician's perception of suitability of the assessment procedures to refine the diagnosis and to target adequate treatment.

SECONDARY OUTCOMES:
Nociceptive pain drivers : Change in Brief Pain Inventory (BPI) scores at 6 weeks | At T2: patient initial visit; T3: +6 weeks after initial visit
  Change in BPI scores measured at T2 and T3 (T3-T2)
Nervous system dysfunction drivers: Change in Pain Detect Questionnaire scores at 6 weeks | At T2: patient initial visit; T3: +6 weeks after initial visit
  Change in Pain Detect Questionnaire scores measured at T2 and T3 (T3-T2)
Nervous system dysfunction drivers: Change in Central Sensitization Index (CSI) scores at 6 weeks | At T2: patient initial visit; T3: +6 weeks after initial visit
  Change in CSI scores measured at T2 and T3 (T3-T2)
Cognitive-emotional drivers: Change in StartBackTool (SBT) scores at 6 weeks | At T2: patient initial visit; T3: +6 weeks after initial visit
  Change in SBT scores measured at T2 and T3 (T3-T2)
Contextual drivers: Change in Orebro Musculoskeletal Pain Screening Questionnaire (OMPSQ) scores at 6 weeks | At T2: patient initial visit; T3: +6 weeks after initial visit
  Change in OMPSQ scores measured at T2 and T3 (T3-T2)

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Tousignant-Laflamme, PhD, Principal Investigator — School of Rehabilitation, University of Sherbrooke
Locations (2):
- Canada (2):
  - Réseau de clinique PhysioExtra, Montreal, Quebec
  - CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Longtin C, Decary S, Cook CE, Martel MO, Lafrenaye S, Carlesso LC, Naye F, Tousignant-Laflamme Y. Optimizing management of low back pain through the pain and disability drivers management model: A feasibility trial. PLoS One. 2021 Jan 20;16(1):e0245689. doi: 10.1371/journal.pone.0245689. eCollection 2021. PMID 33471827
- See also: Website (online resource) linked to the study that will be available to the participating clinicians in order to facilitate their use of the PDDM model — https://pddmmodel.wordpress.com/